CLINICAL TRIAL: NCT02326532
Title: Incorporation of Patient Reported Outcomes Data in the Care of US Veterans With Rheumatoid Arthritis
Acronym: PRO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: North Florida Foundation for Research and Education (Other)
Collaborators: Pfizer (Industry); US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: IRB2014002 18
Record Dates: First submitted 2014-12-09; First posted 2014-12-29 (Estimated); Last update posted 2020-09-09 (Actual); Status verified 2020-09

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis; Veterans
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PRO data utilized (Experimental): PRO data derived from the patient-completed MDHAQ/RAPID3 questionnaire will be collected from this arm and provided to the treating physicians.
  Interventions: Other: PRO data utilized
- PRO data not utilized (Sham Comparator): PRO data derived from the patient-completed MDHAQ/RAPID3 questionnaire will be collected from this arm but will not be provided to the treating physicians.
  Interventions: Other: PRO data not utilized

INTERVENTIONS:
Other: PRO data utilized — Data collected from a patient-completed MDHAQ/RAPID3 questionnaire is provided to the treating physician.
  Arms: PRO data utilized
Other: PRO data not utilized — Data collected from a patient-completed MDHAQ/RAPID3 questionnaire is not provided to the treating physician.
  Arms: PRO data not utilized

SUMMARY:
The overall goal of this proposal is to address barriers to the use of patient reported outcome (PRO) data in the Dept. of Veterans Affairs (VA) health care system.

DETAILED DESCRIPTION:
This is a randomized, controlled, single-blinded study that compares outcome data in patients for whom PRO data either is or is not made available to the treating physician. The question addressed by this proposal is whether patient reported outcome (PRO) data change patient's outcomes. The hypothesis is that the availability of these data in the form of the patient-completed Multidimensional Health Assessment Questionnaire/routine assessment of patient index data (MDHAQ/RAPID3) questionnaire will change patient-centric outcomes such as patient reported well-being, patient satisfaction and medication compliance.

ELIGIBILITY:
Inclusion Criteria:

* US veteran
* Within North Florida/South Georgia (NF/SG) Veterans Integrated Service Network

Exclusion Criteria:

* Outside of service network
* Non-veteran

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 143 (Actual)
Dates: Start 2015-02; Primary Completion 2021-06-01 (Estimated); Study Completion 2021-06-01 (Estimated)

PRIMARY OUTCOMES:
physician/lab-derived instruments of clinical efficacy as measured by DAS28 change and DAS28 remission. | 1 year
  Physician/lab-derived instruments of clinical efficacy as measured by DAS28 change and DAS28 remission.

SECONDARY OUTCOMES:
patient satisfaction | 1 year
  Patient reported satisfaction with medical care. A validated patient satisfaction survey will be collected at study completion with the Leeds Satisfaction Questionnaire.
medication compliance | 1 year
  Degree of medication compliance. Medication compliance will be assessed by the medication possession ratio (MPR) of Methotrexate (MTX), a drug most Rheumatoid Arthritis (RA) patients are prescribed. The VA Pharmacy Benefits Management (PBM) database collects information on medications dispensed and when refills are needed. Thus, a delay in refill will reflect MTX non-compliance. If it MTX is discontinued due to an adverse reaction, it is noted in the electronic medical record. The MPR is calculated as the number of days of prescribed MTX divided by the total number of days of a course.

CONTACTS AND LOCATIONS:
Overall Officials: Michael R Bubb, MD, Principal Investigator — Veterans Health Administration, University of Florida
Locations (1):
- Malcom Randall VAMC, Gainesville, Florida, United States